CLINICAL TRIAL: NCT05008588
Title: Safety and Efficacy of Combined Conditioned Medium With Umbilical Cord Mesenchymal Stem Cells as A Novel Strategy for Acute Stroke Infarct
Brief Title: Combination of Conditioned Medium and Umbilical Cord-Mesenchymal Stem Cells Therapy for Acute Stroke Infarct
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PT. Prodia Stem Cell Indonesia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CT/STROKE/PSI/2021
Record Dates: First submitted 2021-08-01; First posted 2021-08-17 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Ischemic Stroke
Keywords: Ischemic stroke; Mesenchymal Stem Cells; Conditioned Medium; Secretome
MeSH Terms: conditions — Ischemic Stroke | interventions — Culture Media, Conditioned; Secretome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conditioned medium combined with Umbilical cord mesenchymal stem cells treatment (Experimental): Intranasal of 3 cc of conditioned medium each, for 3 days in a row and Intra-parenchymal transplantation of 20x10^6 UC-MSCs
  Interventions: Biological: Conditioned Medium; Biological: Umbilical Cord Mesenchymal Stem Cells
- Umbilical cord mesenchymal stem cells treatment (Experimental): Intra-parenchymal transplantation of 20x10^6 UC-MSCs
  Interventions: Biological: Umbilical Cord Mesenchymal Stem Cells
- Standard treatment (control) (Active Comparator): Neurologic and Neutrophic Drugs
  Interventions: Procedure: Neurologic and Neutrophic Drugs

INTERVENTIONS:
Biological: Conditioned Medium — Intranasal of 3 cc of conditioned medium each, for 3 days in a row
  Other Names: Secretome
  Arms: Conditioned medium combined with Umbilical cord mesenchymal stem cells treatment
Biological: Umbilical Cord Mesenchymal Stem Cells — Intra-parenchymal transplantation of 20x10^6 UC-MSCs
  Other Names: Mesenchymal stromal cells
  Arms: Conditioned medium combined with Umbilical cord mesenchymal stem cells treatment; Umbilical cord mesenchymal stem cells treatment
Procedure: Neurologic and Neutrophic Drugs — Such as clopidogrel, piracetam, citicoline
  Arms: Standard treatment (control)

SUMMARY:
The purpose of this study was to determine the effectiveness of a combination of intranasal conditioned medium (CM) with intraparenchymal umbilical cord mesenchymal stem cells (UC-MSCs) transplantation in acute stroke patients to induce neurogenesis.

DETAILED DESCRIPTION:
This study has 3 arms namely CM and UC-MSCs treatment, UC-MSCs treatment only, and control. The investigator hypothesized that group of CM and UC-MSCs combination is the optimal treatment to induce neurogenesis in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 25-60 years diagnosed with ischemic stroke acute phase
* The patient has had a CT scan/MRI of the brain to assess ischemic territory
* The patient must have an NIH Stroke score of 8-20
* The patient or legal assistant has obtained detailed informed consent regarding the study protocol and agreeing to participate in the study
* Patients with The Glasgow Coma Scale (GCS) score > 8
* Patients with Pt-APTT values within normal limits

Exclusion Criteria:

* Patients with recurrent stroke in the 6 months preceding the episode current stroke
* CT or MRI images show midline shift and bleeding transformation
* Participate in similar studies using CM and/or UC-MSC
* Patients who are immunocompromised and/or who are receiving therapy immunosuppressive
* Patients who cannot have a CT or MRI examination due to their condition
* Patients with impaired renal and hepatic function after the onset of ischemic stroke: Serum Glutamic Oxaloacetic Transaminase (SGOT) and Serum Glutamic Pyruvic Transaminase (SGPT) > 5x the upper limit of normal values and a significant increase in urea-creatinine values
* Patients with a history of malignant tumors or other severe neurologic conditions.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Brain-Derived Neutrophic Factor at one month, 3 months and 6 months after transplantation | Before treatment, one month after treatment, 3 months after treatment, and 6 month after treatment
  Venous blood collection
Change from baseline Vascular endothelial growth factor at one month, 3 months and 6 months after transplantation | Before treatment, one month after treatment, 3 months after treatment, and 6 month after treatment
  Venous blood collection
Change baseline Magnetic Resonance Imaging at 6 month after transplantation | Before treatment, 6 month after transplantation
  To observe the brain development (neurogenesis)

SECONDARY OUTCOMES:
The National Institute of Health Stroke Scale (NIHSS) Scoring | Before treatment, one month after treatment, 3 months after treatment, and 6 month after treatment
  The NIH Stroke Scale (NIHSS) is a 15-item scale that is a well-validated and prognostically important measure of stroke-related neurologic deficits in research and clinical care
modified Rankin Scale (mRS) | Before treatment, one month after treatment, 3 months after treatment, and 6 month after treatment
  The Modified Rankin Scale (mRS) is used to measure the degree of disability in patients who have had a stroke

CONTACTS AND LOCATIONS:
Overall Officials: Rima Haifa, Principal Investigator — Prodia StemCell Indonesia
Locations (2):
- Indonesia (2):
  - Gatot Soebroto Hospital, Jakarta Pusat, DKI Jakarta
  - PT Prodia StemCell Indonesia, Jakarta